CLINICAL TRIAL: NCT00246220
Title: A Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Response Study To Evaluate the Safety And Efficacy Of Prolonged Release OROS Methylphenidate Hydrochloride (18, 36 and 72 mg/Day), With Open-Label Extension, In Adults With Attention Deficit/Hyperactivity Disorder
Brief Title: A Study of the Effectiveness and Safety of Prolonged-release Methylphenidate Hydrochloride in Adult Patients With Attention Deficit/Hyperactivity Disorder.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002479
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention deficit/hyperactivity disorder; methylphenidate; central nervous system stimulants
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate hydrochloride

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of three doses of prolonged-release methylphenidate (a central nervous system (CNS) stimulant) in adult patients with attention deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Stimulant therapy is the mainstay of pharmacologic treatment for attention deficit/hyperactivity disorder (ADHD) in children and adolescents. Methylphenidate is the most commonly prescribed and most frequently studied stimulant medication for children and adolescents with this disorder. It is widely acknowledged in the scientific literature that ADHD often will persist into adulthood. Few large-scale, rigorous studies have been conducted to investigate the effectiveness and safety of stimulant therapy in treating ADHD in adults. This is a multicentre, double-blind, randomised, placebo-controlled, parallel group, dose-response study comparing three doses of prolonged-release methylphenidate (18, 36, and 72 mg once-daily) versus placebo in adult patients with ADHD. The primary efficacy outcome will be the change from baseline to the end of the double-blind phase in the sum of the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated Conners' Adult ADHD Rating Scale (CAARS). Additional measures of effectiveness will include the following scales: CAARS-self report, to rate items pertaining to the patient's behavior/problems; Clinical Global Impression (CGI), to rate the severity of a patient's illness; Sheehan's Disability Scale (SDS), to measure the extent to which a patient's work, social life or leisure activities and home life or family responsibilities are impaired by his/her symptoms; Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q); and the Global Assessment of Effectiveness. Safety and tolerability will be monitored throughout the study. The study hypothesis is that prolonged-release methylphenidate taken once-daily will produce clinically significant improvements compared with placebo on measures of inattention and hyperactivity/impulsivity of the Conners' Adult ADHD Rating Scale in patients with adult ADHD. Prolonged-release methylphenidate 18, 36 or 72 mg oral capsules, or placebo, taken once-daily for 5 weeks. Eligible patients may continue prolonged-release methylphenidate in an open-label extension study for an additional 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD) according to DSM-IV criteria
* ADHD symptoms from childhood to adulthood, with some symptoms present before age 7 years which continue to meet DSM-IV criteria at the time of assessment. (ADHD is not diagnosed if the symptoms are better accounted for by another psychiatric disorder.)

Exclusion Criteria:

* Patients known to be a non-responder to methylphenidate or known to have a child who is a non-responder to methylphenidate
* treated with any methylphenidate-containing medication within 1 month of starting the study
* have any clinically unstable psychiatric condition including, but not limited to the following: acute mood disorder, bipolar disorder, acute obsessive-compulsive disorder, anti-social personality disorder, borderline personality disorder
* family history of schizophrenia or affective psychosis
* patients with motor tics or a history of Tourette's syndrome, or with a substance abuse or dependence disorder, an eating disorder, or mental retardation
* using any medications which may affect the evaluation of study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2005-03; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the sum of the inattention and hyperactivity/impulsivity subscale scores of the investigator-rated Conners' Adult ADHD Rating Scale at the end of the double-blind phase (5 weeks) compared with placebo.

SECONDARY OUTCOMES:
Changes from baseline to the end of treatment in: Conners' Adult ADHD Rating Scale; Clinical Global Impression; Sheehan's Disability Scale; Quality of Life Enjoyment and Satisfaction Questionnaire; and Global Assessment of Effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.

REFERENCES:
- [Result] Medori R, Ramos-Quiroga JA, Casas M, Kooij JJ, Niemela A, Trott GE, Lee E, Buitelaar JK. A randomized, placebo-controlled trial of three fixed dosages of prolonged-release OROS methylphenidate in adults with attention-deficit/hyperactivity disorder. Biol Psychiatry. 2008 May 15;63(10):981-9. doi: 10.1016/j.biopsych.2007.11.008. Epub 2008 Jan 22. PMID 18206857
- [Derived] Buitelaar JK, Sobanski E, Stieglitz RD, Dejonckheere J, Waechter S, Schauble B. Predictors of placebo response in adults with attention-deficit/hyperactivity disorder: data from 2 randomized trials of osmotic-release oral system methylphenidate. J Clin Psychiatry. 2012 Aug;73(8):1097-102. doi: 10.4088/JCP.11m07528. Epub 2012 Jun 12. PMID 22780962
- See also: A Multicentre, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Response Study Evaluating Safety & Efficacy of CONCERTA OROS (18, 36 and 72 mg/day) With Open-Label (OL) Extension in Adults with ADHD — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=378&filename=CR002479_CSR.pdf
- See also: |A Multicentre, Randomized, DB, PCB controlled, Parallel Group, Dose-Response Study to Evaluate Safety and Efficacy of Prolonged Release OROS®methylphenidate (18, 36 and 72 mg/day), With OL Extension, in Adults with ADH — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=378&filename=CR002479_REF1.pdf